CLINICAL TRIAL: NCT00232115
Title: Pimecrolimus Cream 1% in Adult Patients With Perioral Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981CDE15
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2008-01

CONDITIONS: Perioral Dermatitis
Keywords: Perioral Dermatitis, pimecrolimus cream
MeSH Terms: conditions — Dermatitis, Perioral | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus
  Interventions: Drug: Pimecrolimus
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 %
  Other Names: Elidel
  Arms: 1
Drug: Placebo — Vehicle cream (placebo)
  Arms: 2

SUMMARY:
An evaluation of the safety and efficacy of the calcineurin inhibitor, pimecrolimus cream 1%, in adult patients with perioral dermatitis.

This study is not enrolling patients in the United States.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed perioral dermatitis associated or not associated with topical steroid use (the periorbital area may also be involved in addition to the perioral region)
* minimum severity score (PODSI) ≥ 4
* age 18 and older

Exclusion Criteria:

* Ongoing use of the following treatments is NOT allowed after the start of study drug:

Oral tetracyclines, oral erythromycin, oral steroids and oral calcineurin inhibitors. All topical treatments of the face, including steroids, calcineurin inhibitors, metronidazole, tetracyclines, erythromycin and emollients (exception: DAC Basiscreme).

* Systemic immunosuppression
* History of malignancy of any organ system, treated or untreated, within the past 5 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2005-09; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Reduction of the Perioral Dermatitis Severity Index

SECONDARY OUTCOMES:
Time to disease recurrence
Response rates
Patient's quality of life assessment
Patient's disease severity assessment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Nuremberg, Germany

REFERENCES:
- [Derived] Schwarz T, Kreiselmaier I, Bieber T, Thaci D, Simon JC, Meurer M, Werfel T, Zuberbier T, Luger TA, Wollenberg A, Brautigam M. A randomized, double-blind, vehicle-controlled study of 1% pimecrolimus cream in adult patients with perioral dermatitis. J Am Acad Dermatol. 2008 Jul;59(1):34-40. doi: 10.1016/j.jaad.2008.03.043. Epub 2008 May 7. PMID 18462835